CLINICAL TRIAL: NCT01058850
Title: A Phase I Study of Rindopepimut After Conventional Radiation in Children With Diffuse Intrinsic Pontine Gliomas
Brief Title: Phase I Rindopepimut After Conventional Radiation in Children w/ Diffuse Intrinsic Pontine Gliomas
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Resources can be better spent on higher enrolling studies
Sponsor: Paul Graham Fisher (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, Paul Graham Fisher, Professor of Pediatrics, Stanford University
Organization: Stanford University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PEDSBRN0008; SU-01062010-4642 (Other: Stanford University); 1RC2CA148491-01 (NIH)
Record Dates: First submitted 2010-01-27; First posted 2010-01-29 (Estimated); Last update posted 2021-09-27 (Actual); Status verified 2021-09

CONDITIONS: Brain Cancer; Brain Stem Tumors; Pontine Tumors
MeSH Terms: conditions — Brain Neoplasms; Brain Stem Neoplasms | interventions — rindopepimut

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Rindopepimut (EGFRvIII Vaccine, CDX-110) (Experimental)
  Interventions: Biological: Rindopepimut

INTERVENTIONS:
Biological: Rindopepimut — 250 or 500 mcg; intradermal injection
  Other Names: CDX-110, EGFRvIII peptide vaccine

SUMMARY:
This is a research study of patients with diffuse intrinsic pontine gliomas. We hope to learn about the safety and efficacy of treating pediatric diffuse intrinsic pontine glioma patients with the EGFRvIII peptide vaccine after conventional radiation.

ELIGIBILITY:
Inclusion Criteria:

3.1.1 Patients must be at least 3 years of age and ≤ 18 years of age at the time of study enrollment.

3.1.2 Patients must have clinical findings and neuroradiographic findings consistent with diffuse intrinsic pontine glioma. Histologic confirmation of diagnosis is not required for diffuse intrinsic pontine gliomas. A copy of the MRI must be submitted for verification of eligibility.

3.1.3 Patients must have received conventional radiation therapy of total radiation dosage ranging from 5400 to 6000 cGy administered in fractions of 150 to 200 cGy over 6 weeks.

3.1.4 Treatment must start 14 to 28 days after completion of conventional radiation

3.1.5 Patients receiving systemic corticosteroid therapy must be on a tapering or stable low (2 mg twice daily) dose of dexamethasone two weeks after conventional radiation.

3.1.6 Patients life expectancy must be greater or equal to 8 weeks.

3.1.7 Patients must have a performance status (Lansky or Karnofsky) ≥ 50.

3.1.8 Platelet count ≥ 100,000/ mm3.

3.1.9 Hemoglobin ≥ 10 g/dL.

3.1.10 Creatinine ≤ 2.0 mg/dL.

3.1.11 Serum bilirubin ≤ 5.0 mg/dL.

3.1.12 If female, patients of childbearing potential must have a negative serum β-hCG pregnancy test.

3.1.13 Both male and female patients must agree to use hormonal or barrier birth control with spermicidal gel to avoid pregnancy during the study.

3.1.14 The patient and/or their guardian must have the ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria

3.2.1 Prior therapy for diffuse intrinsic pontine glioma, aside from surgery, conventional radiation, and temozolomide.

3.2.2 Use of any experimental drug for any reason within the 60 days prior to treatment.

3.2.3 Active infection requiring treatment.

3.2.4 Known medical condition that, in the opinion of the Investigator, would compromise the patient's ability to participate in the study. This would include chronic active hepatitis infection, known immunosuppressive disease or concurrent neurodegenerative disease.

3.2.5 Known allergy or hypersensitivity to any of the components of the vaccine treatment, including GM-CSF, yeast derived products, or a history of anaphylactic reactions to shellfish proteins.

3.2.6 Pregnant women and women who are breast-feeding.

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 3 (Actual)
Dates: Start 2011-06; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Safety | Monthly until death or until 5years

SECONDARY OUTCOMES:
Overall survival | Monthly until death or until 5years

CONTACTS AND LOCATIONS:
Overall Officials: Paul Graham Fisher, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States